CLINICAL TRIAL: NCT06413446
Title: Evaluation of the Effectiveness of Genicular Block in Postoperative Analgesia in Patients Undergoing Knee Arthroscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Sevil Azazoglu ERBEK, specialist, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024-296
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Knee Pain Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The effectiveness of genicular block in postoperative analgesia management in arthroscopy cases are intended to be evaluated.

DETAILED DESCRIPTION:
Relieving postoperative arthroscopy pain requires multimodal approaches of pain The most common treatment options are nonsteroidal anti-inflammatory drugs (NSAIDs), opioids and local infiltration of anesthetics is used. Due to the side effects of NSAIDs and opioids application of regional analgesia techniques, while providing better analgesia quality.

It can reduce complications . Peripheral blocks such as genicular block, reduce side effects by reducing the use of other analgesics . Pain, it is considered one of the most important factors affecting the quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

Our patients who will be included in the research are patients who underwent arthroscopy under elective conditions.

It consists of volunteers over the age of 18, regardless of gender.

-

Exclusion Criteria:

* Infection in the block area
* Coagulation disorder,
* Known allergy to local anesthetics
* Pregnancy
* Patient with neuropathy
* Uncooperative patient
* The patient who refused to participate in the study
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our patients who will be included in the research are patients who underwent arthroscopy under elective conditions.
  It consists of volunteers over the age of 18, regardless of gender.
  -
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
the perioperative effect of genicular block | 06.10.2024-12.10.2024
  The primary implication of this study is the perioperative effect of genicular block in arthroscopy surgery.
  To show that it has sufficient contribution to multimodal analgesia.

REFERENCES:
- [Background] Singh S, Singh S, Nachimuthu M, Kassim AF, Bhullar AK, Veerakumaran R, Kol GN, Roslan NAM. Effectiveness of Ultrasound-guided versus Anatomical Landmark-guided Genicular Nerve Block to Treat Chronic Knee Osteoarthritis: A Retrospective Cohort Study. Oman Med J. 2023 Sep 28;38(5):e550. doi: 10.5001/omj.2023.103. eCollection 2023 Sep. PMID 38225997
- [Background] Pietrantoni P, Cunat T, Nuevo-Gayoso M, Martin N, Tio M, Basora M, Sastre S, Sala-Blanch X. Ultrasound-guided genicular nerves block: an analgesic alternative to local infiltration analgesia for total knee arthroplasty: A noninferiority, matched cohort study. Eur J Anaesthesiol. 2021 Aug 1;38(Suppl 2):S130-S137. doi: 10.1097/EJA.0000000000001546. PMID 34038916
- [Background] Sahoo RK, Krishna C, Kumar M, Nair AS. Genicular nerve block for postoperative pain relief after total knee replacement. Saudi J Anaesth. 2020 Apr-Jun;14(2):235-237. doi: 10.4103/sja.SJA_611_19. Epub 2020 Mar 5. PMID 32317883